CLINICAL TRIAL: NCT02818036
Title: An fMRI Study of Opioid-related Changes in Neural Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tristen Inagaki (Other)
Responsible Party: Sponsor-Investigator, Tristen Inagaki, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO15010292
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Social Acceptance
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- naltrexone (Experimental): single 50mg dose of naltrexone
  Interventions: Drug: Naltrexone
- sugar pill (Placebo Comparator): single sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone
  Arms: naltrexone
Drug: Placebo
  Arms: sugar pill

SUMMARY:
The purpose of the study is to explore the effect of blocking opioids on affiliation-related neural activity.

ELIGIBILITY:
Inclusion Criteria:

* good health
* between the ages of 18 and 35,
* fluent in English
* right-handed (for the fMRI scan)

Exclusion Criteria:

* Self-reported current or past diagnoses of physical or mental illness.
* Score on the Patient Health Questionnaire (depressive symptoms) above a 13
* Positive urine drug test (for Tetrahydrocannabinol (THC), Opiates, Cocaine, Amphetamine (AMP), and Methamphetamine (mAMP))
* Positive urine pregnancy test
* Use of any prescription medication, except for birth control
* Use of any over-the-counter medications on the day of the fMRI session and 24 hours after the fMRI session
* Self-reported problems with liver functioning, including hepatitis or liver failure
* Difficulty swallowing or taking pills
* BMI greater than 35 or weight greater than 400 lbs
* Claustrophobia
* Nonremovable metal in the body

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2016-08; Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Ross LP, Andreescu C, Inagaki TK. Relationships Between Early Maternal Warmth and Social Connection: A Randomized Clinical Trial With Naltrexone. Psychosom Med. 2021 Oct 1;83(8):924-931. doi: 10.1097/PSY.0000000000000986. PMID 34292204
- [Derived] Inagaki TK, Hazlett LI, Andreescu C. Opioids and social bonding: Effect of naltrexone on feelings of social connection and ventral striatum activity to close others. J Exp Psychol Gen. 2020 Apr;149(4):732-745. doi: 10.1037/xge0000674. Epub 2019 Aug 15. PMID 31414860

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: single 50mg dose of naltrexone
  Naltrexone
- Sugar Pill: single sugar pill
  Placebo
Period: Overall Study
Arm/Group | Naltrexone | Sugar Pill
Started | 42 | 40
Completed | 40 | 40
Not Completed | 2 | 0
Not completed — head did not fit in fMRI scanner headres | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 2 participants were not included from the naltrexone group for final analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Sugar Pill | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.90 (3.49) | 22.88 (3.20) | 22.39 (3.362)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 13 | 19 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 12 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 27 | 23 | 50
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.30 (3.60) | 23.42 (2.61) | 23.86 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Bold Oxygen-level Dependent (BOLD) Activations in Prespecified ROIs
Description: In the MRI scanner, participants read sentences written by people they knew and people they did not know in a block design. Brain activity was measured as BOLD activity in response to reading sentences from known (vs. unknown) people using functional magnetic resonance imaging (FMRI). Based on a priori hypotheses, brain activity was masked to activity in structural regions-of-interest (ROIs) of the ventral striatum (VS) and middle-insula (MI).
Time Frame: approximately one hour after taking study drug
Population: all participants, 3 excluded from sugar pill group (1 for poor registration during preprocessing, 1 for technical error with task presentation, 1 for signal dropout in primary regions of interest)
Measure: Mean (Standard Error); unit: BOLD signal
Arm/Group | Naltrexone | Sugar Pill
Number analyzed (Participants) | 40 | 37
BOLD signal | 0.117 (0.033) | 0.2545 (0.061)
Statistical Analysis 1: Comparison: Naltrexone vs Sugar Pill; Test type: Other — difference in neural activity to social task when taking naltrexone as compared to placebo; p < .01, t-test, 1 sided — a priori threshold for significance was p<.05; degrees of freedom = 75

2. Primary Outcome: Self-reported Feelings of Connection in Response to the Scanner Tasks
Description: feelings of social connection in response to reading sentences from known people (i.e. average of how connected, touched, warm did you feel). Feelings were reported on a scale of 1 (not at all) to 7 (very) such that higher numbers reflect greater feelings of social connection.
  time frame was mistakenly entered as the start of the fMRI scan, but participants reported on their feelings of social connection after the scan. Thus, the outcome measure time frame is reported as two, rather than one, hour after taking the study drug.
Time Frame: approximately two hours after taking study drug
Population: All participants. Ratings from 1 participant in the naltrexone group were misplaced. 1 participant from the sugar pill group did not follow instructions and so ratings were not included in final analyses.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Naltrexone | Sugar Pill
Number analyzed (Participants) | 39 | 39
scores on a scale | 4.576 (.848) | 4.766 (.895)
Statistical Analysis 1: Comparison: Naltrexone vs Sugar Pill; Test type: Other — differences in feelings of social connection between those who took naltrexone and those who took placebo; p = .338, t-test, 2 sided — a priori threshold for statistical significance was p<.05

ADVERSE EVENTS:
Time Frame: Symptoms in response to taking the study drugs were collected approximately three hours after drug administration
Description: Symptoms were collected on a 0 - 4 scale, with 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms, 4 = very severe symptoms.
Arm/Group | Naltrexone | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 30/40 | 20/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=40) | Sugar Pill (N=40)
Nausea (Gastrointestinal disorders) | 6 | 3
Stomach pain (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 28 | 19
Dizziness (Nervous system disorders) | 15 | 4
Headache (Nervous system disorders) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT02818036/Prot_SAP_000.pdf